CLINICAL TRIAL: NCT00498121
Title: The Diagnostic and Prognostic Utility of Procalcitonin (ProCT) for Ventilator-associated Pneumonia (VAP)
Status: Terminated | Type: Observational
Why Stopped: One of the principal investigators has moved to a different institution
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: McGill University Health Center, McGill University Health Center
Other Study IDs: BMA-07-001 (mbasi100)
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator associated pneumonia.; Procalcitonin.
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VAP patient
  Interventions: Device: PROCALCITONIN LEVEL

INTERVENTIONS:
Device: PROCALCITONIN LEVEL — measuring PROCALCITONIN LEVEL

SUMMARY:
Our aim in this study is to investigate the potential role of serum ProCT as an early diagnostic marker and later prognostic indicator for VAP.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP), a bacterial infection that develops after 48 hours or more of intubation, is associated with high morbidity and mortality. Rapid identification of VAP is required to improve survival and to reduce avoidable treatment-associated side effects. Procalcitonin (ProCT), a blood test, is a reasonably specific marker of bacterial infection and its level increases early in sepsis. In this study, a ProCT serum level will be measured in 50 patients with clinically suspected VAP. We aim to show that the ProCT level will be high early in VAP and will stay high in patients with poor prognosis. This will help to address the potential role of ProCT as part of early diagnosis and management of VAP.

ELIGIBILITY:
Inclusion Criteria:

In the preceding 24 h, the appearance of a new opacity or opacities on chest X-ray when compared to previous, and two of the following:

1. white blood cell count > 12 or < 5 x 10^9 cells/L,
2. temperature > 38°C or < 35°C, or
3. purulent secretions.endotracheal samples must be collected by bronchoscope/bronchoalveolar lavage with quantitative culture or endotracheal aspiration with quantitative culture (when available) or qualitative culture from each patient to be enrolled in the study. This is a routine procedure done in every case of suspected VAP and is considered to be the standard of care.

Exclusion Criteria:

1. Known underlying chronic inflammatory condition of the lung (e.g., sarcoidosis, vasculitis)
2. Thyroid cancer patients
3. neutropenia (neutrophils < 0.5 x 10^9 cells/L
4. Concomitant AIDS
5. Solid organ transplantation with severe immunosuppression
6. New Antibiotic use for more than 18 hrs before blood sample collection
7. Severe pancreatitis
8. Attending physician does not agree with enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are intubated or more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Cases with VAP and high ProCT and Cases with Non-VAP and Low ProCT | Retrospective chart review after results are available

CONTACTS AND LOCATIONS:
Overall Officials: Salman A Qureshi, MD,FRCPSC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] Duflo F, Debon R, Monneret G, Bienvenu J, Chassard D, Allaouchiche B. Alveolar and serum procalcitonin: diagnostic and prognostic value in ventilator-associated pneumonia. Anesthesiology. 2002 Jan;96(1):74-9. doi: 10.1097/00000542-200201000-00018. PMID 11753005